CLINICAL TRIAL: NCT00087984
Title: A Phase I/II Study To Examine The Safety, Feasibility, Immunological Response, And Measures Of Clinical Antitumor Activity After Administering Unselected, Autologous, Amplified Tumor Total RNA-Transfected, Dendritic Cell Vaccine (MB-002) To Patients With Metastatic Renal Cell Carcinoma
Brief Title: RNA-Loaded Dendritic Cell Cancer Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MB-002-003
Record Dates: First submitted 2004-07-16; First posted 2004-07-20 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney cancer; Renal cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

ARMS (1):
- MB-002-003 (Experimental)
  Interventions: Biological: MB-002

INTERVENTIONS:
Biological: MB-002 — Dendritic Cell Immunotherapy

SUMMARY:
The purpose of this trial is to examine the safety, feasibility, immunological response, and clinical antitumor activity of administering a dendritic cell vaccine to patients with metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Have a new diagnosis of metastatic renal cell carcinoma;
* Must be at least 18 years or older;
* Have a scheduled unilateral nephrectomy;
* ECOG of 0 or 1;
* Free of brain metastases by CT or MRI;
* Normal renal function in contralateral kidney;
* Male or non-pregnant/non-lactating female on appropriate birth control methods while on study;
* Clinically acceptable screening results.
* No immunosuppressive therapy not limited to corticosteroids (including topical steroids or steroid containing inhalers), azathioprine cyclosporine two months prior to study entry;
* No active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To examine the safety of multiple administrations of MB-002 in patients with newly diagnosed, metastatic renal cell carcinoma. | From registration until disease progression or withdrawal from study
To measure clinical antitumor activity including objective tumor response and an estimate of time to tumor progression (or progression-free interval). | From registration until disease progression or withdrawal from study

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - University of California - Irvine, Orange, California
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- See also: Kidney Cancer Association — http://www.nkca.org